CLINICAL TRIAL: NCT06142331
Title: Investigation of Feasibility and Effectiveness of Home-Based Exercise Programs in Physiotherapy According to Disease Status: A Randomized Controlled Multicenter Study Protocol
Brief Title: Applicability of Home-based Exercise Programs in Physiotherapy
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, doctor, Necmettin Erbakan University
Other Study IDs: ADagbasi002
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Home Exercise
Keywords: home exercise; exercise behavior; exercise compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim: In this study, the types of home-based exercise programs prepared for patients receiving physiotherapy services in different rehabilitation institutions; It is aimed to examine the applicability and effectiveness advantages according to disease status, age, gender, socioeconomic level, education level, confidence in the home program, and functional independence level.

Study type: observational study Research question; To what extent do patients participate in home-based exercise programs?

DETAILED DESCRIPTION:
Background and rationale; It is common to use home exercise programs in organizations that provide physiotherapy services. The home exercise program is specially created by physiotherapists according to the patient's needs and individual characteristics. The prepared program is explained to the patient how to do the exercise at home by various means such as verbal explanation, practical demonstration, giving brochures or video recording. Home program exercises contribute positively to the rehabilitation process by enabling the patient to take an active role in the rehabilitation process and giving the patient personal responsibility. Supporting the treatments given in health institutions with home program exercises increases the effectiveness of the treatment. In addition, preparing a home exercise program is a frequently used method in cases where access to healthcare is difficult due to various reasons.

Aim: In this study, the types of home-based exercise programs prepared for patients receiving physiotherapy services in different rehabilitation institutions; It is aimed to examine the applicability and effectiveness advantages according to disease status, age, gender, socioeconomic level, education level, confidence in the home program, and functional independence level.

Research processes; Participants will first be interviewed face to face and preliminary evaluation data will be obtained before a home exercise program is given.

The patient's gender, age, diagnosis, education level, socioeconomic level, functional dependency level, state anxiety level, fatigue severity scale, and pain level score will be recorded. The type of exercise given and the type of learn home-based exercise will be recorded.

12 days after the routine home exercise program, the final data will be collected by the researchers from the patients face to face or by phone for patients who cannot attend the appointment.

ELIGIBILITY:
Inclusion Criteria:

* Having a clinical problem that causes physiotherapy and rehabilitation treatment
* Being able to understand Turkish

Exclusion Criteria:

* Not wanting to participate in the study
* Having a chronic disease or disability that would prevent the application of the home program.

Max Age: 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population/Sample of the Study: The population of the study consists of patients receiving Physiotherapy and Rehabilitation services in the hospital and rehabilitation center where the health services where the research will be carried out are provided.
  The sample of the research: Consists of 60 volunteer participants under the age of 18 and 177 participants over the age of 18 in the relevant units of three different health institutions, as stated, consisting of women and men. Only 89 female and male volunteer participants over the age of 18 will be included in the study in the physical therapy and rehabilitation unit of our hospital.
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Vizuel Analog Scala, (VAS) | baseline, post-exercise (day 12)
  VAS is an extremely simple, effective and repeatable measurement tool that requires minimal tools to measure both pain intensity and pain relief. It is a 10 cm long ruler drawn horizontally or vertically, starting with "No pain" and ending with "Unbearable pain". The patient is told to make a mark on this line that corresponds to the severity of his pain, intersecting this line. The distance from the lowest VAS level to the patient's mark is measured with a ruler to obtain a numerical index of the patient's pain intensity in cm or mm.

SECONDARY OUTCOMES:
Fatigue Severity Scale, (FSS) | baseline, post-exercise (day 12)
  Fatigue Severity Scale is a scale with proven validity and reliability. FSS is shown as the best example among one-dimensional scales. The person indicates how much he or she agrees with each item by choosing a number from 1 to 7. 1 indicates that it does not agree at all, 7 indicates that it completely agrees. The score range of the scale, which consists of a total of 9 questions, is 9-63. A score of 36 or higher indicates severe fatigue.

OTHER OUTCOMES:
Functional independence measure, (FIM) | baseline, post-exercise (day 12)
  FIM analyzes two different aspects of disability, namely motor and cognitive functions. It consists of 6 functional parts: self-care, sphincter control, mobility, locomotion, communication and social perception. In the FIM, a total of 18 activities are evaluated for functional independence using a 7-point scale for each. The highest score that can be obtained is 126. The Turkish version of FIM was used in our study.
State Anxiety Scale | baseline, post-exercise (day 12)
  The state anxiety inventory was developed to measure a person's anxiety at a certain moment. The state anxiety inventory, consisting of 20 items, is a scale that determines how the individual feels at a certain moment and condition. The emotions or behaviors expressed in the state anxiety inventory items are answered by marking one of the options: (1) not at all, (2) a little, (3) a lot, (4) completely, according to the degree of intensity. There are 10 inverted expressions in the inventory.
Functional Independence Measure for Children (WeeFIM) | baseline, post-exercise (day 12)
  It contains a total of 18 items in 6 areas: self-care, sphincter control, transfers, movement, communication, social and cognitive. Each item in these areas is scored from 1 to 7, depending on whether the person receives help while performing the function, whether it is done on time, or whether an assistive device is required. When the given task is done completely with assistance, it is evaluated as 1, and when it is done completely independently, at the appropriate time and safely, it is evaluated as 7.
Gross Motor Function Classification System (GMFCS) | baseline, post-exercise (day 12)
  It is a 5-level classification system. Children with cerebral palsy under the age of 12 are divided into five levels based on gross motor functions such as self-initiated movements, sitting, and walking. Level 1: Walks independently. There are limitations in advanced gross motor skills. Level 2: walks without aids. There are limitations when walking in public. Level 3: Walks with an assistive device. There are limitations when walking in public. Level 4: It has a limitation. It is mobile by itself. Moves or uses a wheelchair (TS) in public. Level 5: mobilization is severely limited, although assistive technologies are used.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Altuntaş Yılmaz, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim JY, Lee MK, Lee DH, Kang DW, Min JH, Lee JW, Chu SH, Cho MS, Kim NK, Jeon JY. Effects of a 12-week home-based exercise program on quality of life, psychological health, and the level of physical activity in colorectal cancer survivors: a randomized controlled trial. Support Care Cancer. 2019 Aug;27(8):2933-2940. doi: 10.1007/s00520-018-4588-0. Epub 2018 Dec 18. PMID 30564936